CLINICAL TRIAL: NCT01048047
Title: Effects of Aliskiren/Amlodipine Versus Amlodipine Monotherapy on Ankle-foot Volume in Hypertensive Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Pavia (Other)
Responsible Party: Roberto Fogari, University of Pavia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UNIPV001DIM2009; EudraCT 2009 (Registry Identifier: EudraCT 2009-016479-30)
Record Dates: First submitted 2010-01-12; First posted 2010-01-13 (Estimated); Last update posted 2010-01-13 (Estimated); Status verified 2009-11

CONDITIONS: Hypertension
Keywords: aliskiren; amlodipine; hypertension; ankle-foot volume; mild and moderate hypertension
MeSH Terms: conditions — Hypertension; Lymphoma, Follicular | interventions — aliskiren; Amlodipine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- aliskiren/amlodipine (Experimental): aliskiren, 300 mg/amlodipine 10 mg
  Interventions: Drug: aliskiren/amlodipine
- amlodipine (Active Comparator): amlodipine 10 mg
  Interventions: Drug: aliskiren/amlodipine

INTERVENTIONS:
Drug: aliskiren/amlodipine — aliskiren 300 mg /amlodipine 10 mg

SUMMARY:
Comparison between the effect of aliskiren/amlodipine combination with amlodipine monotherapy on ankle-foot volume in hypertensive patients. It will be enrolled male or female outpatients, aged 18-65 years.

ELIGIBILITY:
Inclusion Criteria:

* diastolic blood pressure > 95 mmHg and < 110 mmHg
* systolic blood pressure > 140 mmHg and < 180 mmHg
* no amlodipine therapy for the previous 6 months

Exclusion Criteria:

* diastolic blood pressure > 110 mmHg and or
* systolic blood pressure > 180 mmHg
* secondary hypertension
* heart failure
* diabetes mellitus
* liver or kidney diseases

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2009-11; Primary Completion 2009-12 (Estimated); Study Completion 2010-03 (Estimated)

PRIMARY OUTCOMES:
Blood pressure, heart rate, ankle-foot volume | At baseline, at the end of the wash-out period, after 2, 4, and 8 weeks

SECONDARY OUTCOMES:
Blood pressure and heart rate in sitting and standing position | At baseline, at the end of the wash-out period, after 2, 4, and 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Roberto Fogari, MD, Principal Investigator — University of Pavia
Locations (1):
- University of Pavia, Pavia, Italy